CLINICAL TRIAL: NCT00890734
Title: A Double-blind, Placebo-controlled Study to Assess Pharmacodynamic and Clinical Efficacy of CYT003-QbG10 in Patients With Persistent Allergic Asthma Bronchial
Brief Title: CYT003-QbG10 for Treatment of Allergic Asthma Bronchial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT003-QbG10 11
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Allergic Bronchial Asthma
MeSH Terms: interventions — CYT003-QbG10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CYT003-QbG10
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CYT003-QbG10 — subcutaneous injection
  Arms: 1
Drug: Placebo — subcutaneous injection
  Arms: 2

SUMMARY:
The purpose of the study is to test whether treatment with CYT003-QbG10 can improve asthma symptoms in patients with allergic bronchial asthma. The active treatment will be compared against placebo.

ELIGIBILITY:
Inclusion Criteria:

* Persistent allergic asthma bronchial requiring long-term treatment with inhaled corticosteroids
* Further criteria as defined in the study protocol

Exclusion Criteria:

* Use of oral corticosteroids within past 3 months
* Hospitalization for asthma exacerbation within past 6 months
* Uncontrolled asthma
* Contraindication to any study test or procedure
* Further criteria as defined in the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Markers for inflammation and asthma | 1-3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cytos Investigator Sites, Luebeck, Berlin, Wiesbaden, Rodgau, Eisenach, Germany

REFERENCES:
- [Derived] Beeh KM, Kanniess F, Wagner F, Schilder C, Naudts I, Hammann-Haenni A, Willers J, Stocker H, Mueller P, Bachmann MF, Renner WA. The novel TLR-9 agonist QbG10 shows clinical efficacy in persistent allergic asthma. J Allergy Clin Immunol. 2013 Mar;131(3):866-74. doi: 10.1016/j.jaci.2012.12.1561. Epub 2013 Feb 4. PMID 23384679